CLINICAL TRIAL: NCT07372547
Title: Effect of Voiding Position (Standing in the Shower vs. Sitting) on Post-Void Residual Urine Volume (PVR) After Removal of Urinary Catheter in Women Following Benign Vaginal Gynecologic Surgery: A Double-Blind Randomized Controlled Trial
Brief Title: Effect of Voiding Position (Standing in the Shower vs. Sitting) on Post-Void Residual Urine Volume (PVR) After Removal of Urinary Catheter in Women Following Benign Vaginal Gynecologic Surgery
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assuta Ashdod Hospital (Other)
Responsible Party: Principal Investigator, Elad Preuss, Principal Investigator, Gynaecologist, Assuta Ashdod Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: AAA-0147-25
Record Dates: First submitted 2026-01-04; First posted 2026-01-28 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Post-void Residual Volume; Recatheterization; Pain; UTI; Urinary Retention
MeSH Terms: conditions — Pain; Urinary Retention

STUDY DESIGN:
Who Masked: Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Voiding position - Standing in the shower (Other): After removal of urine catheterization, during first micturation, the patient will stand in the shower with the water on her vulvar area
  Interventions: Behavioral: Voiding position - Standing in the shower
- Voiding position - Sitting on the toilet (Other): After the removal of urine catheter for the first micturation - the patient will sit on the toilet
  Interventions: Behavioral: Voiding position - Sitting on the toilet

INTERVENTIONS:
Behavioral: Voiding position - Standing in the shower — After the removal of urine catheter, for the first micturation the woman will stand in the shower with the water on her vulvar area
  Arms: Voiding position - Standing in the shower
Behavioral: Voiding position - Sitting on the toilet — After the removal of urine catheter, for the first micturation the women will sit on the toiled
  Arms: Voiding position - Sitting on the toilet

SUMMARY:
The goal of this clinical trial is to learn if voiding in a standing position in the shower, rather than sitting on a toilet, may reduce pain associated with the act of voiding, thereby facilitating micturition and decreasing both post-void residual volume and the risk of subsequent urinary retention in women that underwent benign vaginal surgeries.

ELIGIBILITY:
Inclusion Criteria:

* Adult women (≥18 years old).
* Undergoing benign vaginal gynecologic surgery with indwelling catheter during surgery.
* No bladder injury during surgery.
* Ability and willingness to consent.
* No known neurological or urinary conditions affecting voiding.
* No active urinary tract infection at time of catheter removal.

Exclusion Criteria:

* Bladder injury during surgery.
* Neurological disease affecting bladder function.
* Active urinary tract infection.
* Inability to void either standing in shower or sitting (depending on randomization).

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 100 (Estimated)
Dates: Start 2026-01-20 (Estimated); Primary Completion 2028-01-20 (Estimated); Study Completion 2028-01-20 (Estimated)

PRIMARY OUTCOMES:
Post-void residual volume>150 CC | The following 7 days after surgery
  after the first void following catheter removal

SECONDARY OUTCOMES:
Success rate of voiding trial | The following 7 days after surgery
  no need for recatheterization
Pain during micturition | The following 7 days after surgery
  Pain during micturition, using The Visual Analogue Scale (VAS) 0-10. O means no pain, 10 means worst pain imaginable.
UTI | The following 7 days after surgery
  in the 7 days following the surgery
Urinary retention | The following 7 days after surgery
  REST>150 ml
Post-void residual volume | The following 7 days after surgery
  in ml

CONTACTS AND LOCATIONS:
Locations (1):
- Assuta Ashdod Hospital, Ashdod, Israel